### VA RESEARCH CONSENT FORM


Subject Name: SSN: Date:

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: Lori L. Davis, MD VAMC: Tuscaloosa
Co- Investigators: Patricia Pilkinton, MD Version Date: August 9, 2021

#### INTRODUCTION

We are asking you to volunteer to take part in a research study at the Tuscaloosa Veterans Affairs Medical Center (TVAMC). It is important that you read and understand the information on this form. The sponsor (financial source) for this study is Pharmacotherapies for Alcohol and Substance Abuse (PASA) Consortium.

#### **BACKGROUND AND PURPOSE**

Currently four medications (disulfiram, oral and long-acting injectable naltrexone, and acamprosate) are FDA-approved to treat alcohol use disorder (AUD) and two medications (sertraline and paroxetine) FDA-approved to treat post-traumatic stress disorder (PTSD). Despite a growing body of research in this area, there are no medications shown to be clearly effective when heavy drinking and PTSD co-occur. This study addresses the need for new and effective treatments. The purpose of this study is to evaluate how well the combination of sublingual buprenorphine (SL-BUP; Subutex) combined with extended-release injectable naltrexone (XR-NTX; Vivitrol) works in the treatment of co-occurring AUD and PTSD. In addition, we are also trying to learn what happens to a person's physical responses to unexpected sounds, lights, images, and air puff while viewing computer images of neutral, trauma-related, and alcohol-related topics. You are possibly eligible for this study because you may have recent heavy alcohol use and symptoms of PTSD. Your study participation will last approximately 15 weeks. You will be one of approximately 90 to 135 people across three medical centers to participate in this study.

### STUDY PROCEDURES

Baseline Assessments: After signing the informed consent, you will meet with someone from the research team to be screened for the study (lasting several hours over 1 to 14 days), which includes answering questions about your mental health conditions, drinking patterns and PTSD symptoms, filling out pen-and-paper surveys about your alcohol use, PTSD symptoms, depression symptoms, life activities, and tendencies to be impulsive, and getting your blood drawn for basic laboratory tests, which includes a urine drug screen in the research clinic. At the screening and baseline visits, you will be assessed for signs and symptoms of withdrawal from alcohol. If you have signs such as unstable pulse, blood pressure, or sweating or symptoms such as tremor, nausea, vomiting, agitation, feeling crawling sensations on skin, or hallucinations, we may recommend a referral to mental health provider for alcohol detoxification treatment. The results of the urine drug screen remain in the research records and do not go into your VA records. You will also be asked to blow into a breathalyzer to test for alcohol level and these results will be kept in the research records, but the results will not be entered into your VA records unless there is a serious safety issue that requires medical intervention. If the drug screen is positive for any drugs (except marijuana) and/or you have a breathalyzer level > 0.02 or positive blood alcohol level. the appointment will be canceled, and you will not be paid for this appointment. In addition, we are also trying to learn what happens to a person's physical responses to unexpected sounds, lights, images, and air puff while viewing computer images of neutral, trauma-related, and alcohol-related topics. We may

IRB Use Only:

VA FORM

JAN 1990 **10-1086** Revised: September 28, 2015

### VA RESEARCH CONSENT FORM


Subject Name: SSN: Date:

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: Lori L. Davis, MD VAMC: Tuscaloosa Co- Investigators: Patricia Pilkinton, MD Version Date: August 9, 2021

be able to reschedule your appointment for a later date. You may continue some allowed medications that are prescribed for PTSD, but you cannot take other psychiatric medication or medication used to treat AUD during the study.

<u>Study Medications</u>: At the baseline visit, the research medication provider orders the study medication and the VA pharmacy dispenses the study medication or placebo medication according to the computer-generated assignment to one of two treatments in a random order (i.e. like flipping a coin). You will be taking the assigned treatment during the next 12 weeks (i.e. the dose will not change); however, you will not know which one of the three treatments you are assigned from the following list:

- SL-BUP 2mg and XR-NTX 380mg, or
- SL-placebo and XR-placebo; You have 1 in 2 chances of being on placebo.

XR-NTX or XR-placebo given by injection in your gluteal muscle (buttocks) in the research clinic by a trained research nurse or medical doctor on the day it is dispensed from the pharmacy and every 28-days on week 4 and week 8 of the study. You will receive the first injection of XR-NTX or XR-placebo in the research clinic and remain in the clinic under the supervision of the research team for approximately 1 hour after the 1<sup>st</sup> dose is administered.

SL-BUP or SL-placebo is started on the next day, taken sublingually (in other words, place and hold the table under your tongue until it dissolves) and is taken daily at the same time every day. If you miss a dose, you should take the next dose as soon as possible. You will be given enough pills needed to allow one pill per day for each day to last until the date of your next scheduled visit. It is important that you keep your appointments so that you do not run out of medication. Bring any remaining medication back to the next research appointment.

Do not share your study drug with others, keep study drug secured (in your possession or locked up), keep study drug out of reach of children and pets. Bring any unused study drug back to the pharmacy when you return.

If for any reason there is study medication that will go permanently unused, the research coordinator will give you a Take-Away Medication Recovery System tamper-resistant envelope and you will place the unused medication in this envelope and put in a US postal service mailbox to be sent to a pharmacy destruction service.

<u>Follow-Up Visits:</u> You will be evaluated by phone or video telehealth at week 1, 2, 6, and 8; however, you return to the research clinic for in-person assessments on weeks 4, 8, and 12. If you prefer all visits to be conducted in person, we will honor your preference. The research coordinator will also contact you by telephone (t) during the weeks between face-to-face visits to remind you of the next office visit and to check on adherence to the study medication and if there have been any serious adverse events.

The investigators and a research coordinator will meet with you to provide ongoing reinforcement of your commitment to the study participants. The study medication provider will emphasize the need to properly adhere to prescribed study medication or to call to revise the treatments if side effects occur or therapeutic effects are lost. The face-to-face assessments will include your answering questions about

IRB Use Only:

VA FORM

JAN 1990 **10-1086** Revised: September 28, 2015

### VA RESEARCH CONSENT FORM


Subject Name: \_\_\_\_\_ Date: \_\_\_

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: Lori L. Davis, MD VAMC: Tuscaloosa
Co- Investigators: Patricia Pilkinton, MD Version Date: August 9, 2021

your mental health conditions, drinking patterns and PTSD symptoms, filling out pen-and-paper surveys about your alcohol use, PTSD symptoms, depression symptoms, life activities, and a urine drug screen in the clinic. The results of the urine drug screen remain in the research records and do not go into your VA records. You will also be asked to blow into a breathalyzer to test for alcohol level at all research visits and these results will be kept in the research records, but the results will not be entered into your VA records unless there is a serious safety issue that requires medical intervention. At week 8 and 12, you will also have your blood drawn for an alcohol-related blood lab test.

While every attempt is made to retain you in the study on medication for the full 12 weeks, you may discontinue medication at any point and remain in the study for assessments through week 12. If you exit prior to week 8, all procedures for week 8 are completed. If you exit after week 8 but prior to week 12, all week-12 procedures are completed. The investigator may discontinue your study participation without your consent for reasons of safety or your nonadherence to the study procedures.

At week 12, the study medications are discontinued, and all week 12 assessments are completed. A member of the research team will call you a few days later to make sure you have not had any problems with stopping the study medication. At week 12, you will be referred back to your previous or newly assigned long-term PTSD provider for follow-up and continued treatment. At week 14, you will be assessed for discontinuation or withdrawal side effects and resolution or emergence of adverse events, either in-person visit or by video telehealth visit.

For women of childbearing potential: Since it is unknown whether the study drug may have bad effects on an unborn child and should not be taken during pregnancy, it is necessary that a pregnancy test be done during screening and during follow-up. If you are a woman of child-bearing potential, you will be asked to have a urine pregnancy test in the clinic to make sure that you are not pregnant. You agree to use contraceptives and take precautions against becoming pregnant during this study.

Because this is a new combination of drugs, we do not know all side effects. You should contact Dr. Pilkinton at 205-554-2000 ext. 1-2944 or Dr. Lori Davis at ext. 1-3819 if you have any side effects.

We cannot guarantee that you will be able to continue receiving this medication after this study is over. Naltrexone is currently on VA formularies and you may have access to this medication from your clinic provider. Although SL-BUP is on VA formulary, it is not currently indicated for AUD or PTSD.

#### While in the study, your responsibilities include:

Take the study medication as instructed and return unused study drug to the research team. Keep your study appointments and let the investigator know if you are having problems. If you miss an appointment, please contact the research coordinator to reschedule. Keep your study drug in a safe place for your use only and away from children or pets. Do not take part in any other research project without talking it over with the investigator. Do not take additional or new medication without talking it over with the investigator.

Psychophysiological Assessments (OPTIONAL): At baseline (two days), week 2 (one day), and week 8 (two days), you may choose to undergo a psychophysiological assessment that will take place

IRB Use Only:

VA FORM

JAN 1990 **10-1086** Revised: September 28, 2015

### VA RESEARCH CONSENT FORM


Subject Name: \_\_\_\_\_ Date: \_

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: Lori L. Davis, MD VAMC: Tuscaloosa
Co- Investigators: Patricia Pilkinton, MD Version Date: August 9, 2021

over two days (lasting approximately 1 hour and 10 minutes on day one and 30 minutes on day two). You will be asked to complete several tasks where we will monitor your physical reactions to lights, sounds, and images. We will measure how strong your eyes blink, the amount of sweat on your hands, and changes in your heart rate and breathing throughout the tasks. You will receive additional compensation for participating in this part of the study.

We will measure these responses by placing electrodes (tiny metal discs with wires attached to them) on your skin which will send information to a computer. Before placing the electrodes, a member of the research team will clean the following areas with alcohol and/or a gritty gel: the left forearm, right collarbone, and just below your right eye. The electrodes will then be placed below your eye, arm, collarbone, and fingers.

Next, a brief hearing test will be conducted. During the first task, you will be seated in a sound-proof booth and given instructions for the task. Next, you will hear sounds through headphones while lights in the booth switch between "on" and "off". You may be startled when you hear these sounds and you may blink your eyes. The electrodes will allow us to measure how strongly you blink your eyes. During the second task, you will see a series of shapes on a computer screen and hear sounds through the headphones. There will be some mildly uncomfortable events, including short puffs of air pointed toward your neck, but these will not be painful. When each shape appears, you will be asked to press a button indicating what you think the shape means in the context of the task. You will also view a computer-generated virtual reality environment that includes victim-reported contexts associated with assault (e.g. barracks, latrines, rear seat of a vehicle). These contexts do not recreate the traumatic events that may have led to the development of PTSD. You will also repeat the task while viewing images related to alcohol cues. During the 2nd day, we will administer another task like those described above, although the 2nd day is much shorter duration.

#### PHOTOGRAPHY, VIDEO AND/OR AUDIO RECORDING FOR RESEARCH PURPOSES

During the assessment of your PTSD symptoms and alcohol use, the interview will be audio-recorded for purposes of making sure that the person conducting the interview is adhering to the questions and making the assessment of your symptom severity according to our study plan. This recording will be listened to by a study monitor and your information will be kept confidential. This recording will not be shared with your providers, the public, or other members of the research team.

#### POSSIBLE RISKS OR DISCOMFORTS

Any procedure has possible risks and discomforts. The procedures in this study may cause all, some, or none of the risks or side effects listed. Rare or unexpected risks also may occur. Risks of the usual health care you receive are not risks of the research and are not listed in this consent form. If you have any questions about the risks of your usual care, you should talk with your health care providers.

<u>Questionnaires/interview-based assessments</u> may bring up painful emotions, such as sadness, worry, or increased anxiety or upsetting memories, such as trauma-related events or periods of heavy alcohol use. You are free to take breaks or to not answer a question. To minimize the risk, the person

IRB Use Only:

VA FORM

JAN 1990 **10-1086** Revised: September 28, 2015

### VA RESEARCH CONSENT FORM


Subject Name: SSN: Date:

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: <u>Lori L. Davis, MD</u> VAMC: <u>Tuscaloosa</u>
Co- Investigators: <u>Patricia Pilkinton, MD</u> Version Date: <u>August 9, 2021</u>

doing the interview is trained to ask the questions with respect and dignity and allow you to express how you feel without causing blame or shame.

<u>Venipuncture (blood draw)</u>: It is unlikely, but for some people the blood draw(s) may cause discomfort, pain, bruising, <u>and</u> rarely, fainting, or infection. These procedures are done only by skilled and experienced laboratory or research personnel to reduce the risk of any negative reactions.

**Sublingual buprenorphine:** Sublingual buprenorphine (SL-BUP) is FDA-indicated for the treatment of opioid dependence. SL-BUP is a Schedule III narcotic under the Controlled Substances Act. The use of SL-BUP in a non-opioid dependent population has a risk of misuse or abuse. However, to essentially eliminate the potential for misuse, dependency, and withdrawal, SL-BUP is combined with XR-NTX, a medication that blocks the brain receptor involved in euphoric properties of buprenorphine. Adverse events most commonly observed during clinical trials and post-marketing experience for SL-BUP compared to placebo are headache (29% vs 22%), nausea (14% vs 11%), vomiting, hyperhidrosis, constipation (8% vs 3%), signs and symptoms of withdrawal (18% vs 37%, i.e. greater in placebo group), insomnia (21% vs 16%), and pain (18% vs 19%). The doses used in this study are lower and may yield fewer side effects. Since the SL-BUP dosing is low, there is only a very low risk (% unknown) of having symptoms of upset stomach, headache, or sweating for a few days after you discontinue the medication. If this happens, the doctors or nurse practitioner can give you non-controlled medication to help reduce symptoms.

Significant respiratory depression and death have occurred in association with buprenorphine, particularly when taken by the intravenous (IV) route in combination with benzodiazepines or other CNS depressants (including alcohol). Many, but not all post-marketing reports regarding coma and death associated with the concomitant use of buprenorphine and benzodiazepines involved misuse by self-injection. To minimize these risks, you are not allowed to take benzodiazepines (i.e., Ativan, Valium, Xanax, Klonopin, etc.) and anti-seizure medications during the study.

Extended-release naltrexone: Side effects of XR-NTX that led to more discontinuation of treatment compared to placebo include the following: pain, tenderness, induration or pruritus at the site of the injection (3%), nausea (2%), headache (1%), and suicide-related events (0.3%). Other known non-serious side effects that differ from placebo include nausea (29% vs 11%), vomiting (12% vs 6%), diarrhea (13% vs 10%), abdominal pain (11% vs 8%), injection site reactions (65% vs 50%), arthralgia/arthritis (9% vs 5%), muscle cramps (5% vs 1%), rash (6% vs 4%), headache (21% vs 18%) dizziness (13% vs 4%), somnolence/sedation (5% vs 1%), and appetite decrease (11% vs 3%). XR-NTX has the capacity to cause liver injury when given in excessive doses (five-fold times the recommended dose). Thus, XR-NTX does not appear to be a risk to the liver at the recommended doses used in this study. Since naltrexone gradually leaves your body over time, there is no risk of withdrawal symptoms after you discontinue the medication.

In a situation when analgesia (i.e. sedative for surgery) may be required, consideration should be given to regional analgesia, conscious sedation with a benzodiazepine, use of non-opioid analgesics, or general anesthesia. If opioid analgesia is required, the amount of opioid needed may be greater than usual, and the resulting respiratory depression may be deeper and more prolonged. In this case, a

IRB Use Only:

VA FORM

JAN 1990 10-1086

Revised: September 28, 2015

Tuscaloosa VAMC IRB Effective Date:

### VA RESEARCH CONSENT FORM


Subject Name: \_\_\_\_\_ Date: \_

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: Lori L. Davis, MD VAMC: Tuscaloosa Co- Investigators: Patricia Pilkinton, MD Version Date: August 9, 2021

rapidly-acting opioid analgesic that minimizes the duration of respiratory depression is preferred. XR-NTX can also diminish the benefit from opioid-containing cough, cold, and antidiarrheal preparations. These warning are standard when treating patients with XR-NTX and a safety card will be provided to you for you to carry in your wallet or purse in case of emergency.

<u>Combination of SL-BUP and XR-NTX:</u> The occurrence of side effects may be slightly more frequent (22% of people taking the combination compared to 18% for XR-NTX) but the type of side effect does not change when the two medications are used in combination. The combination of these medications may reduce the desire to use more SL-BUP than otherwise prescribed.

<u>Caution:</u> Do not drive or operating hazardous machinery until you are reasonably certain that treatment does not adversely affect your ability to engage in such activities. If you experience a medical emergency, informed the emergency team that you may be on these medications so that they know how to treat you.

The risks of complications during pregnancy or congenital problems with this drug combination is not fully known, although much is known about each medication separately. There is no evidence that either medication affects reproductive risks after discontinuation. Similarly, there is no evidence that either medication affects male reproductive risks.

There may be unknown risks or discomforts involved. Study staff will update you in a timely way on any new information that may affect your decision to stay in the study.

<u>Psychophysiology tasks:</u> It is somewhat likely that scrubbing your skin in the places where the monitor pads are placed may cause redness or mild swelling. The noise level you will hear during the session should not result in any discomfort but may be mildly annoying. You may find the air blasts, darkness, small room, or virtual reality contexts somewhat annoying or uncomfortable. To reduce this risk, the tasks are performed at your own pace and in a private clinic office. You may ask for the session to be stopped immediately if you are uncomfortable or distressed. The decibel levels and duration of the auditory stimuli are not sufficient to cause any damage to the ear.

#### POTENTIAL BENEFITS

We cannot promise that you will get any benefits from taking part in this study. XR-NTX is FDA approved for the treatment of alcohol dependence, as well as for the prevention of relapse to opioid dependence, following opioid detoxification. Thus, XR-NTX may directly benefit you in this study and help you reduce or stop the use of alcohol. Reducing alcohol use may also be a factor in reduction of PTSD symptoms and conversely, reduced PTSD symptoms may lower your tendency to self-medicate with alcohol. Another benefit of the study is that knowledge to be gained can help guide treatment for patients with comorbid AUD and PTSD in the future.

#### OTHER TREATMENT AVAILABLE

If you do not wish to participate in this study, you may continue in your present treatment or you may be referred to a mental health clinic or PTSD clinic for additional treatment.\_

IRB Use Only:

VA FORM

JAN 1990 10-1086

Revised: September 28, 2015

Tuscaloosa VAMC IRB Effective Date:

### VA RESEARCH CONSENT FORM


Subject Name: \_\_\_\_\_ Date: \_

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: Lori L. Davis, MD VAMC: Tuscaloosa
Co- Investigators: Patricia Pilkinton, MD Version Date: August 9, 2021

Four medications (disulfiram, oral and long-acting injectable naltrexone, and acamprosate) are FDA—approved to treat alcohol use disorder (AUD). If you would like to try these medications without being in the study, you need to be referred to or stay in treatment for a mental health provider. There are two medications (sertraline and paroxetine) FDA-approved to treat post-traumatic stress disorder (PTSD). If you are already taking these medications, you may continue them at a steady dose during the study.

You may also seek counseling as treatment for AUD and PTSD. During the study, you can participate in supportive counseling for PTSD or 12-step programs for alcohol problems. However, you are not allowed to participate in cognitive behavioral or prolonged exposure therapies during the study. If you want to participate in these treatments, you may do so either before or after your study participation.

### **CONFIDENTIALITY**

Taking part in this study will involve collecting confidential information about you, including your name, address, phone number, and the surveys that you complete during the study. If you decide to participate, your identity will be protected. Individuals who participate will be assigned a study ID number, which will be kept on a secure network server that complies with all VA Data Security regulations. In order to participate in the study, you will be asked for your contact information (telephone and address) and the name of alternate contact if we are unable to locate you. This information will be protected in the following ways: the information collected will be kept in locked files and on computers protected with passwords. Electronic data will be access-restricted to approved research study staff and will be stored on a secure network server that complies with all VA Data Security Regulations. Information collected for this study will be stored such that only research personnel with permission to see the data will have access to it. Any hard copies will be kept in a locked file cabinet that only study staff will have access to. A copy of this consent form will be place in your medical record.

To minimize breach or invasion of privacy, records that have personal identifiers (i.e., clinical records or source documents) are stored in a locked cabinet behind a locked door. Only the research team and clinical staff assigned to your care have access to non-anonymous research records. Research case report forms do not contain personal identifiers and are labeled with a study i.d. number. Files that link your name with screening and randomization numbers are maintained in a secure location either on VA server or in a locked file within a locked office in the research clinic.

The study findings will be reported in the aggregate, meaning that information about you will be combined with information from other people taking part in the study. Any talks or written papers about this study will not identify you by name, by recognizable photograph, or by any other means without your specific consent. If results of this study are reported in medical journals or at meetings, you will not be identified by name, by recognizable photograph, or by any other means without your specific consent. No presentation or publication of the study results will refer to you individually.

All study participant research data, which is for the purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the PASA Consortium Data Coordinating Center (DCC). This will not include your contact or directly identifying information. Rather, you and your research data will only be identified by a unique study identification number. The study data entry and study management systems used by the clinical site and PASA Consortium Management will be secured and

IRB Use Only:

VA FORM

JAN 1990 10-1086

Revised: September 28, 2015

Tuscaloosa VAMC IRB Effective Date:

### VA RESEARCH CONSENT FORM


| Subject Name: | SSN: | Date: |
|---------------|------|-------|

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: Lori L. Davis, MD VAMC: Tuscaloosa
Co- Investigators: Patricia Pilkinton, MD Version Date: August 9, 2021

password protected. In addition, if you experience a serious adverse event, the investigators will make a report that does not contain your name or identity to the PASA Consortium and to Alkermes (the manufacturer of XR-NTX), as well as to the local IRB; however, the dates and details about the serious event will be provides to the PASA Consortium and to Alkermes. In addition, any pregnancy that occurs during the study and the outcome of the pregnancy will also be reported to PASA Consortium and to Alkermes.

Additionally, as this study is funded by the Department of Defense, a version of the data set will ultimately be made available to the research community (which includes both scientific and consumer advocacy communities) and to the public at large. Those datasets do not include any identifying information. This data will be used for other research studies in the future. If you do not agree that your data be used in future studies, you will NOT be able to participate in this study.

The investigators will treat your identity with professional standards of confidentiality. Your medical records will be maintained according to this medical center's confidentiality requirements. However, there are times when we might have to show your records to other people who have oversight of the study. For example, the Food and Drug Administration, other federal oversight agencies, representatives of the PASA Consortium, members of our Data and Safety Management Board, the Medical Monitor (Dr. Tom Kosten), members of the Government Steering Committee, and/or the VA Institutional Review Board (IRB) may inspect your records, particularly if there is a safety issue. The Research Compliance Officer (RCO) will review this form and may review your other records. A person responsible for monitoring the PTSD and alcohol interview will listen to an audio recording of the interview, but you will not be identified by name or anything other than study i.d. number.

The investigator's research records for this study will be maintained according to the disposition instructions by the National Achieves and Records Administrations and are published in VHA's Records Control Schedule (RCS) 10-1, in accordance with the new VHA's Records Control Schedule 10-1 (RCS) policies for the Office of Research and Development; section 7.6. For a study such as this one, the instructions state that the PI may destroy research records 6 years after the end of the fiscal year after completion of the research project, but the investigator may retain longer if needed.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a> as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

A federal **Certificate of Confidentiality**, which protects your records against subpoena, has been approved for this study. Exceptions to confidentiality are those required by law and include suspicion of child abuse, elder abuse, and threat of imminent action on suicidal or homicidal ideation. The Certificate of Confidentiality cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of Federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an

IRB Use Only:

VA FORM

JAN 1990 **10-1086** Revised: September 28, 2015

### VA RESEARCH CONSENT FORM


Subject Name: \_\_\_\_\_ Date: \_\_\_\_\_

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: Lori L. Davis, MD VAMC: Tuscaloosa Co- Investigators: Patricia Pilkinton, MD Version Date: August 9, 2021

insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

#### WITHDRAWAL FROM STUDY

You are not required to take part in this study: your participation is entirely voluntary. You can refuse to participate at this time, or you can withdraw from the study at any time without penalty or loss of benefits to which you are otherwise entitled. Regarding information already collected prior to your withdrawal, the investigator may continue to review the data already collected for the study but cannot collect further information. Results from laboratory specimens already used cannot be withdrawn.

Your treatment, payment, enrollment or eligibility for benefits will not be affected if you choose not to take part in the study. If you decide to withdraw from this study, you should contact Lori Davis, MD or Patricia Pilkinton, MD. Discontinuation will in no way affect the quality of care you receive now, or in the future, at this institution or your right to participate in other studies. The investigator or your doctor may also withdraw you without your consent, for medical or administrative reasons, in a study that has not ended. Any significant new findings that develop during the research study that, in the opinion of the investigator, may affect your willingness to continue to participate will be provided to you ASAP.

### COST TO YOU FOR PARTICIPATION IN RESEARCH

There will be no costs to you for any of the treatment or testing done as part of this study. Eligibility for medical care is based upon the usual VA eligibility policy and is not guaranteed by participation in a research study. Depending on your veteran status, you might have to pay co-payments for medical care and services provided by VA. Alkermes and Tonix has donated some of the medication used in this study, so there will be no cost to you for the study medication. There is no guarantee that the medicines you will receive during this study will be continued after the study is completed.

#### PAYMENT FOR PARTICIPATION IN THE RESEARCH

You will be paid according to the table below to offset out of pocket expenses such as parking, travel, childcare, missed work, etc. Your personal information will be provided to the Tuscaloosa Research and Education Advancement Corporation so that they can make a check out or give you a cash card to pay you within 30 days of your visit. If you live >50 miles away, you will be given a \$25 gas card for each office visit that attend in which you (or other) drives a vehicle to the appointment. You will NOT be paid for the screening visit if you test positive for any drugs (except marijuana) and/or have a positive blood alcohol level or breathalyzer alcohol level > 0.02. You will only get paid for the visits that you attend.

| Schedule of Payments for Completed Visits | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen | Baseline | 1 | 2 | Т | 4 | Т | 6 | Т | 8 | Т | 10 | Т | 12 | Т | 14 |
| Payments (\$) | 25 | 75 | 25 | 25 | | 75 | | 25 | | 75 | | 25 | | 50 | | 25 |

If you opt in to participate in the psychophysiologic assessments, you will get paid \$25 per day (total of \$125 for all 5 days).

IRB Use Only:

VA FORM

JAN 1990 **10-1086** Revised: September 28, 2015

### VA RESEARCH CONSENT FORM


Subject Name: \_\_\_\_\_ Date: \_

Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD

Principal Investigator: <u>Lori L. Davis, MD</u> VAMC: <u>Tuscaloosa</u>
Co- Investigators: <u>Patricia Pilkinton, MD</u> Version Date: <u>August 9, 2021</u>

**Please note:** if you receive research payments of \$600 or more in each calendar year, an IRS Form 1099 will be sent to you and you will need to report this as income when filing your income tax return. The Form 1099 will include your full social security number.

#### INJURY COMPENSATION CLAUSE

This research project has been approved by the Tuscaloosa VA Institutional Review Board and R&D Committee, and it is being supervised by one or more VA employees. Every reasonable safety measure will be used to protect your well-being. If you are injured as a result of taking part in this study, the Tuscaloosa VA Medical Center will provide you with the necessary medical treatment at no cost to you unless the injury was due to your not following the study procedures. This care is governed by Federal regulations and VA policy. Non-emergency, non-VA Treatment requires prior authorization. Financial compensation is not available for such things as lost wages, disability or discomfort due to an injury. The Department of Veterans Affairs does not normally provide any other form of compensation for injury. You have not released this institution from liability for negligence.

#### **NEW FINDINGS**

You and your physician will be informed if any important discoveries are made during this study which may affect you, your condition, or your willingness to participate in this study. Information obtained in this study which, in the opinion of the investigator(s), suggests that you may be at significant risk of harm to yourself or others will be reportable to a third party in the interest of protecting the rights and welfare of those at potential risk.

#### **QUESTIONS**

If you have questions, concerns or complaints about your rights as a study participant, you may contact the Research Compliance Officer, at (205) 554-2000, ext. 3200 or the Institutional Review Board (IRB) Administrator who will have the IRB member subject representative contact you. The IRB Administrator can be reached at (205) 554-2000, ext. 3674 (Tuscaloosa VA Patients). If the IRB Administrator cannot be reached, contact the IRB Clerical Assistant at (205) 554-2000, ext. 2536 and she will direct your call to an IRB member.

If you have questions regarding this study or the procedures, if you have unexpected reactions, or if you are injured and become ill as a result of participation in this study, please call Dr. Patricia Pilkinton at (205) 554-2000, ext. 2944 or 1-888-269-3045, ext. 2944 (toll free); or Dr. Lori Davis at (205) 554-3819. You may also call the Tuscaloosa VA operator at (205) 554-2000 or 1-888-269-3045 (toll free) and have the operator page Dr. Patricia Pilkinton or Dr. Lori Davis.

If you are unable to reach Dr. Pilkinton or Dr. Davis and need immediate medical assistance for research-related injury, please call the Tuscaloosa VAMC hospital operator at 205-554-2000 or 1-888-269-3045 and ask for the Triage Nurse to obtain advice or ask to speak with the psychiatrist or medical officer on duty.

If for any reason, you experience suicidality, please call 911 or the Suicide Prevention Hotline at 1-800-273-8255, or the TVAMC Suicide Prevention Coordinator at (205) 554-2000 ext. 3235.

IRB Use Only:

VA FORM

JAN 1990 **10-1086** Revised: September 28, 2015

# VA RESEARCH CONSENT FORM

| -1 | | (Page 11 | 1 of 12) |
|---|---|---|---|
| Subject Name: | SSN: | | Date: |
| Title of Study: KOR Antagonism for | the Treatment o | f Alcohol Use Diso | rder and Comorbid PTSD |
| Principal Investigator: Lori L. I | | | IC: <u>Tuscaloosa</u> |
| Co- Investigators: <u>Patricia Pilki</u> | nton, MD | Version Date: | August 9, 2021 |
| AGREEMENT TO PARTICIPATE IN TH | E RESEARCH S | STUDY | |
| RESEARCH SUBJECTS' RIGHTS: You | u have read or l | nave had read to | you all of the above. |
| One of the above listed investigators or a and answered all your questions. You h the study. You have been told of other chance to ask questions and obtain answered. | ave been told of<br>choices of treatm | the risks or discon | nforts and possible benefits of |
| You voluntarily consent to participate in to or loss of rights to which you are entitled study. You may withdraw from this study which you are entitled. | this study, and yo<br>. Your will receiv | e contact informat | tion regarding the research |
| The results of this study may be published | ed but your recor | ds will not be reve | aled unless required by law. |
| In case there are medical problems or if Patricia Pilkinton at (205) 554-2000, ext. at (205) 554-3819. You may also call the (toll free) and have the operator page Dr | 2944 or 1-888-2<br>e Tuscaloosa VA | 69-3045, ext. 2944<br>operator at (205) | 4 (toll free); or Dr. Lori Davis<br>554-2000 or 1-888-269-3045 |
| If any medical problems occur in connec accordance with your eligibility. | tion with this stud | dy, the VA will prov | vide emergency care in |
| You will receive a copy of this consent a your medical record if applicable. | fter you sign it. A | A copy of this signe | ed consent will also be put in |
| I prefer to opt in or opt out _<br>Initials li | of the ps | sychophysiologic | assessments. |
| I agree to participate in this research s | tudy as has been | explained in this do | ocument. |
| Participant's Name | Participant's | s Signature | <br>Date |
| · | | | |

IRB Use Only:

VA FORM

JAN 1990 10-1086 Revised: September 28, 2015

> Tuscaloosa VAMC IRB Effective Date:

# VA RESEARCH CONSENT FORM **VA** Department of Veterans Affairs  SSN: **Subject Name:** Date: Title of Study: KOR Antagonism for the Treatment of Alcohol Use Disorder and Comorbid PTSD Principal Investigator: Lori L. Davis, MD VAMC: Tuscaloosa Co- Investigators: Patricia Pilkinton, MD Version Date: August 9, 2021 Signature of person obtaining consent Name of person obtaining consent Date

IRB Use Only:

VA FORM

JAN 1990 10-1086 Revised: September 28, 2015